CLINICAL TRIAL: NCT02425774
Title: Anti-inflammatory Effect of Pre-operative Stimulation of the Cholinergic Anti-Inflammatory Pathway: A Potential New Therapeutical Intervention for Postoperative Ileus
Brief Title: Anti-inflammatory Effect of Pre-operative Stimulation of the Cholinergic Anti-Inflammatory Pathway
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: S56328
Record Dates: First submitted 2015-02-24; First posted 2015-04-24 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Ileus
Keywords: Prucalopride; Vagus Nerve Stimulation; Postoperative Ileus
MeSH Terms: interventions — Vagus Nerve Stimulation; prucalopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham stimulation + Placebo (Placebo Comparator): * no stimulation
  * 1 placebo tablet at two different timepoints before surgery
  Interventions: Procedure: Sham stimulation; Drug: Placebo
- Vagus stimulation + placebo (Active Comparator): * Stimulation at the beginning and the end of the surgery
  * 1 placebo tablet at two different timepoints before surgery
  Interventions: Procedure: Vagus stimulation; Drug: Placebo
- Prucalopride + sham stimulation (Active Comparator): * 1 prucalopride tablet at two different timepoints before surgery
  * no stimulation
  Interventions: Procedure: Sham stimulation; Drug: Prucalopride

INTERVENTIONS:
Procedure: Vagus stimulation
  Arms: Vagus stimulation + placebo
Procedure: Sham stimulation
  Arms: Prucalopride + sham stimulation; Sham stimulation + Placebo
Drug: Prucalopride
  Arms: Prucalopride + sham stimulation
Drug: Placebo
  Arms: Sham stimulation + Placebo; Vagus stimulation + placebo

SUMMARY:
Hypothesis:

Prucalopride can mimic electrical stimulation of the abdominal vagus nerve and has an anti-inflammatory effect.

Aims:

In the present pilot study, the investigators want to evaluate the anti-inflammatory effect of prucalopride. The following aims are formulated:

1. to show that prucalopride has a similar inflammatory effect as abdominal vagus nerve stimulation (VNS)
2. to evaluate whether prucalopride leads to accelerated post-operative recovery

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing partial or full resection of the pancreas due to a benign or malignant tumor

Exclusion Criteria:

* adjuvant radiotherapy
* evident intra-abdominal inflammation (diagnosed by imaging and/or laboratory results, including an abscess or cholecystitis)
* chronic pancreatitis
* pancreatic polypeptide producing endocrine tumor
* American Society of Anesthesiologists physical-health status classification (ASA-PS)>3
* Poorly regulated diabetes (>200 mg/dl (=11 mmol/l))

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Levels of pro-inflammatory cytokines in intestinal tissue, serum, peritoneal lavage and supernatant of stimulated whole blood | From the date of surgery until the date of lab analysis (up to 6 months)

SECONDARY OUTCOMES:
Time to first flatus | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to tolerance of oral food intake | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to tolerance of oral food intake AND first defecation | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to first defecation | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Gastrointestinal symptoms (nausea, pain, vomiting, bloating) | From the date of surgery until the date of discharge from the hospital (on average 14 days)
Time to discharge from the hospital | From the date of surgery until the date of discharge from the hospital (on average 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Boeckxstaens, M.D., Principal Investigator — Catholic University Leuven
Locations (1):
- University hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Kalff JC, Buchholz BM, Eskandari MK, Hierholzer C, Schraut WH, Simmons RL, Bauer AJ. Biphasic response to gut manipulation and temporal correlation of cellular infiltrates and muscle dysfunction in rat. Surgery. 1999 Sep;126(3):498-509. PMID 10486602
- [Background] Kalff JC, Schraut WH, Simmons RL, Bauer AJ. Surgical manipulation of the gut elicits an intestinal muscularis inflammatory response resulting in postsurgical ileus. Ann Surg. 1998 Nov;228(5):652-63. doi: 10.1097/00000658-199811000-00004. PMID 9833803
- [Derived] Stakenborg N, Labeeuw E, Gomez-Pinilla PJ, De Schepper S, Aerts R, Goverse G, Farro G, Appeltans I, Meroni E, Stakenborg M, Viola MF, Gonzalez-Dominguez E, Bosmans G, Alpizar YA, Wolthuis A, D'Hoore A, Van Beek K, Verheijden S, Verhaegen M, Derua R, Waelkens E, Moretti M, Gotti C, Augustijns P, Talavera K, Vanden Berghe P, Matteoli G, Boeckxstaens GE. Preoperative administration of the 5-HT4 receptor agonist prucalopride reduces intestinal inflammation and shortens postoperative ileus via cholinergic enteric neurons. Gut. 2019 Aug;68(8):1406-1416. doi: 10.1136/gutjnl-2018-317263. Epub 2018 Nov 24. PMID 30472681